CLINICAL TRIAL: NCT06345846
Title: Tilt, Centration and Stability of Secondary Intraocular Lenses With no Capsular Support
Brief Title: Stability of Secondary Intraocular Lenses With no Capsular Support
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Secondary IOL
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Cataract
Keywords: Secondary IOL; Stability
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFIOL (Experimental): Patients with an implanted IFIOL
  Interventions: Device: IFIOL
- SFIOL (Experimental): Patients with an implanted SFIOL
  Interventions: Device: SFIOL

INTERVENTIONS:
Device: IFIOL — Implanted IFIOL
  Arms: IFIOL
Device: SFIOL — Implanted SFIOL
  Arms: SFIOL

SUMMARY:
Assessment and differences in the centration, tilt and wobble of two secondary IOLs without capsular support.

DETAILED DESCRIPTION:
Acquired or congenital weakness of the zonules, either as part of a pseudoexfoliation syndrome (PEX), high myopia, past ocular trauma, post vitreoretinal surgery, and recurrent uveitis are the most common reasons for implantation of a secondary intraocular lenses (IOL) after cataract surgery. There are several techniques available to implant a secondary IOL in eyes with inadequate capsular support. Some of the most common techniques are the placement of a chamber angle-supported anterior chamber IOL (ACIOL), an iris-fixated IOL (IFIOL) and several different possibilities of scleral fixation of the IOL (SFIOL).

While those methods have all been found to show high safety and efficiency, there are certain procedure-specific limitations. One approach to sutureless implantation of a SFIOL is the "double needle flanged technique" described by Yamane et al. When using this technique, there is no need for extensive scleral incisions or distinct scleral manipulation, however, it may be challenging for the surgeon and may lead to complications such as "iris-optic-capture".

Past studies found no significant difference of postoperative best corrected visual acuity or rate of complications when comparing the three mentioned techniques, therefore, up to now choice of implantation and fixation technique lies with the surgeon's preferences and abilities. However, all three techniques have their drawbacks.

Hence, the aim of this study is to assess the centration, tilt, and wobble of secondary IOLs (comparing an IFIOL and a SFIOL) without capsular support.

ELIGIBILITY:
Inclusion Criteria:

* Secondary IOL implantation performed at the Hanusch Hospital
* IFIOL or SFIOL implanted
* Older than 21 years
* Written informed consent prior to recruitment

Exclusion Criteria:

* Concurrent participation in another drug or device clinical investigation
* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Centration of the IOL | 24 months
  Centration of the IOL will be measured in mm using a Purkinjemeter

SECONDARY OUTCOMES:
Tilt of the IOL | 24 months
  Tilt of the IOL will be measured in degrees using a Purkinjemeter

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Krankenhaus
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided